CLINICAL TRIAL: NCT02897011
Title: Effect of Two-week Discontinuation of Methotrexate on Efficacy of Seasonal Influenza Vaccination in Patients With Rheumatoid Arthritis: A Randomized Clinical Trial
Brief Title: 2-week dc of MTX and Influenza Vaccination in RA
Acronym: 2 wk MTX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Bong Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNUH-IMJ-003
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Rheumatoid Arthritis; Influenza; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid; Influenza, Human | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: MTX continue (Sham Comparator): Group will continue MTX after vaccination
  Interventions: Drug: Methotrexate
- Group 2: MTX hold (Experimental): will hold MTX for 2 weeks after vaccination
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate

SUMMARY:
To investigate whether a transient discontinuation of methotrexate MTX for 2 weeks improves the vaccination response to a seasonal influenza.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic systemic inflammatory disease that affects the joints as the main target of the inflammation. Patients with RA require chronic treatment with disease modifying antirheumatic drugs (DMARDs) including methotrexate (MTX), which constitutes the mainstay of treatment. Underlying immune dysfunction and the additional immune suppression associated with treatment render patients with RA more susceptible to infection. Thus, vaccination of the preventive diseases is crucial and recommended in all patients unless contraindicated.

However, low dose of glucocorticoids, conventional DMARDs and biological DMARDs including tumor necrosis factor inhibitors have been reported to substantially decrease vaccine response (4); MTX has been reported to be associated with a decreased response to seasonal influenza vaccination by up to 15%.

To optimize a vaccine response, vaccination should be administrated before the treatment with immunesuppressive medications is initiated. However, most patients with RA are already on stable dose of MTX at the time of when vaccinations. To improve the vaccine response, a short term discontinuation of MTX could be considered. In a prior study, we discovered that a temporary discontinuation of MTX for 4 weeks during peri-vaccination period tended to be associated with an improved response to vaccination with trivalent influenza vaccination (Figure 1). It remains to be defined whether MTX discontinuation for shorter period increases the vaccination efficacy while minimizing the RA flare rate.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 19 years and < 65 years of age at time of consent
* Have a diagnosis of RA per ACR criteria
* Must understand and voluntarily sign an informed consent form including writing consent for data protection
* Stable doses of methotrexate over the preceding 6 weeks

Exclusion Criteria:

* Pregnant or lactating females
* Previous anaphylactic response to vaccine components or to egg.
* Acute infection with T >38°C at the time of vaccination
* History of Guillain-Barre syndrome or demyelinating syndromes
* Previous vaccination with any live vaccine 4 weeks before or any inactivated vaccine 2 weeks before the study
* Blood transfusion within 6 months
* Active rheumatoid arthritis necessitating a recent change in the drug regimen
* Any other rheumatic disease such as systemic lupus erythematosus, mixed connective tissue disease, dermatomyositis/polymyositis, and vasculitis except for secondary Sjogren's disease
* Any condition including laboratory abnormality which places the subject at unacceptable risk
* Subjects who decline to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of satisfactory vaccine response | 4 weeks
  Proportion of satisfactory vaccine response that is defined as ≥ 4-fold increase in post-vaccination titer in ≥ 2 of 4 influenza strains

SECONDARY OUTCOMES:
Proportion of patients who have ≥ 4-fold increase in post-vaccination titer in ≥ 3 of 4 influenza strains | 4 weeks
Proportion of seroprotection for each strain | 4 weeks
Change from baseline in titer (in GMT) for each strain | 4 weeks
Change from baseline in DAS28-4 (CRP) at 4 weeks after vaccination | 4 weeks
Proportion of patients who experience increase in disease activity | 4 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Seoul National Univ. Bundang Hospital, Bundang, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Seoul
  - SMG-SNU Boramae Medical Center, Seoul, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park JK, Choi Y, Winthrop KL, Song YW, Lee EB. Optimal time between the last methotrexate administration and seasonal influenza vaccination in rheumatoid arthritis: post hoc analysis of a randomised clinical trial. Ann Rheum Dis. 2019 Sep;78(9):1283-1284. doi: 10.1136/annrheumdis-2019-215187. Epub 2019 Mar 23. No abstract available. PMID 30904830
- [Derived] Park JK, Lee YJ, Shin K, Ha YJ, Lee EY, Song YW, Choi Y, Winthrop KL, Lee EB. Impact of temporary methotrexate discontinuation for 2 weeks on immunogenicity of seasonal influenza vaccination in patients with rheumatoid arthritis: a randomised clinical trial. Ann Rheum Dis. 2018 Jun;77(6):898-904. doi: 10.1136/annrheumdis-2018-213222. Epub 2018 Mar 23. PMID 29572291